CLINICAL TRIAL: NCT00501605
Title: A Phase I Single Centre 2-part Open Study to Assess the Safety and Tolerability of AZD2171 Following Single and Multiple Oral Doses in Patients With Advanced Solid Malignant Tumors and Liver Metastases
Brief Title: Phase I Study With AZD2171 in Patients With Advanced Solid Malignant Tumors and Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00001
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Advanced Solid Tumor; Liver Metastases
Keywords: Phase I; AZD2171; advanced solid tumors
MeSH Terms: interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZD2171

SUMMARY:
Single centre recruiting approximately 80 patients who are given a rising single, followed by multiple, ascending oral dose of AZD2171, assessing the safety and tolerability of AZD2171 in patients with solid tumors and metastatic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male/female, 18 yr or over
* WHO status 0-2
* Refractory advanced solid tumor

Exclusion Criteria:

* Radiotherapy within 4 weeks of starting AZD2171 treatment
* Low haemoglobin level
* Low platelet or neutrophil counts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2003-02; Primary Completion 2005-04 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
primary objective is to evaluate the safety and tolerability of ascending single&multiple oral doses of AZD2171 by assessment of AEs,BP,HR,RR,ECG,clinical chemistry,haematology,urinalysis incl 24hr collection for protein&creatinine and physical exam.

SECONDARY OUTCOMES:
PK,assess the effects of AZD2171 on surrogate markets of activity and to make a preliminary assessment of anti-tumor activity by measurement of tumor response and time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Nick Botwood, BSc, MBBS, MRCP, MFPM, Study Director — AstraZeneca; J. Drevs, PD, Principal Investigator — Klinik fur.Internistische Onkologie
Locations (1):
- Research Site, Freiburg im Breisgau, Germany